CLINICAL TRIAL: NCT06180850
Title: Building Lipedema Research Resources
Acronym: BRR
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aaron W. Aday, MD, MSc, Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 212427
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lipedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — A standard blood draw will be acquired. Up to 60 mL will be acquired in a 1-time visit.
  Urine collection procedures.
  Tissue punch biopsy taken from the following locations:
  The peri-umbilical region, right upper inner-thigh, left upper inner-thigh
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants with lipedema
- Controls: Participants without lipedema

SUMMARY:
Lipedema is a disease marked by subcutaneous adipose tissue accumulation in the lower extremities of females that is accompanied by somatic pain and edema. Importantly, lipedema is commonly misdiagnosed as obesity, although it's estimated to affect a high 11% of women. Clinical diagnosis of lipedema requires specialized training not widely available at most major medical centers, and there remains a substantial need for objective tools to distinguish lipedema from obesity. There is a critical need to define specific molecular markers of disease in circulation or at the tissue-level. The purpose of this study is to create, manage, and characterize an innovative lipedema biorepository. The goal of the biorepository will be to better understand disease mechanisms of lipedema and to define specific molecular markers of disease in circulation or at the tissue-level. The long-term purpose of our studies are to help with prevention and early management of lipedema.

ELIGIBILITY:
Inclusion Criteria:

* Participants with or without lipedema
* Age range = 18-80 years
* Participants with lipedema have a formal diagnosis by a physician using criteria in Appendix A of protocol
* Female

Exclusion Criteria: Volunteers in the lipedema or control group will be excluded with the following:

* Pregnant or breast-feeding
* Taking any anticoagulation or antiplatelet therapy other than aspirin (up to 100 mg daily)
* Active infection anywhere in the body, or open wound on the lower-extremities or at locations for ultrasound, bioimpedance, and tissue dielectric measurements
* Battery-operated device implanted that cannot be removed for ultrasound, DXA scan, bioimpedance, and tissue dielectric measurements
* Primary lymphedema
* Uncontrolled diabetes, renal disease, thyroid disease, or hypertension
* Hormone dysregulation or another significant clinical condition affecting hormone status as confirmed by clinical co-investigators
* Bone metastases
* Contrast imaging scan in the previous 7 days
* Nuclear medicine scan in previous 3 days
* Lumbar spine fusion
* Weigh more than 500 lb (226.8 kg)

Also excluded are subjects incapable of giving informed written consent:

* Subjects who have an inability to communicate with the researcher for any reason
* Subjects who are non-English speaking who cannot communicate through a translator, or if a translator is not available
* Subjects who cannot adhere to the experimental protocols for any reason
* Subjects who have limited mental ability to give informed consent due to mental disability, confusion, or psychiatric disorders
* Prisoners

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with or without lipedema
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
We will measure plasma concentrations of CD8A. | 1 day
We will measure plasma concentrations of high-sensitivity C-reactive protein. | 1 day

SECONDARY OUTCOMES:
We will measure the 6-minute walk test. | 1 day
We will measure the four-meter gait speed test. | 1 day
We will measure the hand grip strength test. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided